CLINICAL TRIAL: NCT01580189
Title: Effects of Whole Milk Versus Whey Protein Supplementation With Resistance Exercise on Body Composition, Muscle Hypertrophy and Strength Changes in Healthy Individuals
Brief Title: Whole Milk Versus Whey Protein Supplement and Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: B2011:068
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Muscle Development
Keywords: Lean tissue; Strength condition; Protein; Amino Acid
MeSH Terms: interventions — Whey Proteins; Milk; Sugars; maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Milk (Active Comparator): Chocolate milk compared to protein supplement
  Interventions: Dietary Supplement: Whey protein
- Whey protein (Active Comparator): Whey protein compared to milk
  Interventions: Dietary Supplement: Chocolate milk
- Sugar (Placebo Comparator): Maltodextrin compared to treatments
  Interventions: Dietary Supplement: Sugar

INTERVENTIONS:
Dietary Supplement: Whey protein — 18g protein, immediately after training, 9 weeks
  Other Names: protein supplement
  Arms: Milk
Dietary Supplement: Chocolate milk — 500ml chocolate milk, immediately after training, 9 weeks
  Other Names: Milk
  Arms: Whey protein
Dietary Supplement: Sugar — 55-65g maltodextrin solution, immediately after training, 9 weeks
  Other Names: Maltodextrin
  Arms: Sugar

SUMMARY:
The purpose of the study is to examine the effects of consuming protein supplement (whey) compared to whole milk immediately after bouts of resistance training on muscular strength and body composition.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* currently working out at least 3 times per week

Exclusion Criteria:

* taken any ergogenic aid/sport supplements in the last 2 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Body composition | 9 weeks
  DEXA for assessment of fat and lean tissue
Strength | 9 weeks
  1RM tests to assess changes in strength on various sport resistant exercise equipment

SECONDARY OUTCOMES:
Blood amino acid | 9 weeks
  Assessment of plasma amino acid profile at baseline, mid and end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Semone B Myrie, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada